CLINICAL TRIAL: NCT06564337
Title: A Prospective Clinical Trial Evaluating Outcomes of Surveyed Zirconia Crowns on Removable Partial Denture Abutment Teeth
Brief Title: A Prospective Clinical Trial Evaluating Outcomes of Surveyed Zirconia Crowns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neena DSouza (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor-Investigator, Neena DSouza, Co-Investigator, University of Toronto
Organization: University of Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00042791
Record Dates: First submitted 2024-08-18; First posted 2024-08-21 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Removable Partial Denture; Dental Crown
Keywords: removable partial denture abutment; monolithic zirconia crown survival; surveyed zirconia crown

STUDY DESIGN:
Intervention Model Description: Research data on the survival of zirconia crowns as RPD abutments is limited although anecdotally these are being used regularly by dentists in clinical practice. To our knowledge a clinical trial evaluating the outcomes of surveyed monolithic zirconia crowns as RPD abutments has not been investigated previously. We propose to evaluate the outcomes of surveyed zirconia crowns as RPD abutments in a prospective trial and compare the survival, biological and technical complications with alternative materials historically used for surveyed crowns.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients recruited for intervention (Experimental): A combination of 3Y-TZP and 5Y-TZP (IPS e.max ZirCAD Prime, Ivoclar AG) with a flexural strength of 1200MPa will be utilized for the crowns. Tooth preparation will include occlusal reduction of 1.0 to 1.2mm and rounded line angles for the rest seats within the zirconia crown and buccal and lingual reduction of 1 to 1.5mm to allow for adequate buccal and lingual contour to accommodate retentive clasp arms and minor connectors. Impressions for zirconia crowns will be made with polyvinyl siloxane on a full arch custom tray. After clinical verification crowns will be cemented with resin or resin modified glass ionomer cement
  Interventions: Device: Surveyed zirconia crown

INTERVENTIONS:
Device: Surveyed zirconia crown — Patient recruitment will be from the patient population that presents to the undergraduate dental clinic requiring removable dental prosthesis (RPD) to replace missing teeth. Selection of abutment teeth for zirconia surveyed crowns will be similar to that currently utilized when selecting RPD abutments to be restored with either porcelain fused to metal or full metal surveyed crowns for tissue and tooth supported RPD's.

SUMMARY:
Zirconia has shown to be a suitable substitute for metal ceramic crowns when comparing survival, biological and technical complications. Evidence demonstrating the outcomes of surveyed zirconia crowns on removable partial denture abutments is unavailable. Zirconia as a substitute for metal ceramic is being currently used for fabricating surveyed crowns although quantitative data evaluating its efficacy is sparse. The purpose of this prospective clinical trial is to evaluate clinical outcomes when zirconia is used as a full coverage restoration on removable partial denture abutments. The study will be designed as a 3-5 year prospective observational trial in the University of Toronto undergraduate clinic in a controlled environment. Outcomes measures will include survival, biological and technical complications. Descriptive statistics will be used to summarize patient characteristics and outcomes and for categorical variables frequency and percentages will be reported. A level of significance 0.05 will be used for inferential analysis, with p-values < 0.05 reported as statistically significant. It is expected that zirconia will demonstrate similar outcomes to traditional metal ceramic surveyed crowns.

DETAILED DESCRIPTION:
Research data on the survival of zirconia crowns as RPD abutments is limited although anecdotally these are being used regularly by dentists in clinical practice. To our knowledge a clinical trial evaluating the outcomes of surveyed monolithic zirconia crowns as RPD abutments has not been investigated previously. We propose to evaluate the outcomes of surveyed zirconia crowns as RPD abutments in a prospective trial and compare the survival, biological and technical complications with alternative materials historically used for surveyed crowns.

Aims of Project

1. To evaluate biological and technical complications of surveyed zirconia crowns on RPD abutments for 3- 5 years following insertion.
2. To evaluate survival of surveyed zirconia crowns for 3- 5 years following insertion.

Materials and Methods

Research Design and Overview: The study will be designed as a 3-5 year prospective observational trial in the University of Toronto undergraduate clinic in a controlled environment where procedures are standardized for case selection and execution. All patients requiring surveyed crowns in the academic years 2024 and 2025 will be approached to participate in the trial. Patients will be recalled every year for 3-5 years following insertion and a check list will be used to assess the pre insertion and outcome variables. Clinical coordinators supervising students and clinical examiners performing outcome assessments at yearly follow up will be trained and their measurements calibrated for inter and intra observer variability to ensure uniformity. The research proposal will be submitted to the University Research Oversight and Compliance office for ethics approval.

Participant recruitment: Patient recruitment will be from the patient population that presents to the undergraduate dental clinic requiring removable dental prosthesis to replace missing teeth. Selection of abutment teeth for zirconia surveyed crowns will be similar to that currently utilized when selecting abutment teeth to be restored with either porcelain fused to metal or full metal surveyed crowns for tissue and tooth supported cast removable partial dentures. These will include but are not limited to abutment teeth which require full coverage due to large restorations, posterior endodontically treated teeth with inadequate marginal ridge support and abutment teeth which require axial modification for retentive and or stability elements of the denture.

Sample Size Calculation: This is an exploratory study and will include all patients in the undergraduate clinic requiring surveyed crowns. We expect approximately 25-50 surveyed crowns per year, based on numerical data for metal ceramic surveyed crowns done in previous years.

Methods: To avoid the inherent fractures associated with veneered zirconia surveyed crowns, monolithic zirconia a combination of 3Y-TZP and 5Y-TZP (IPS e.max ZirCAD Prime, Ivoclar AG) with a flexural strength of 1200MPa will be utilized. Tooth preparation will include occlusal reduction of 1.0 to 1.5mm and rounded line angles for fabrication of the rest seats within the zirconia crown and buccal and lingual reduction of 1 to 1.5mm to allow for adequate buccal and lingual contour to accommodate retentive clasp arms and minor connectors within the crown. Impressions for zirconia crowns will be made with polyvinyl siloxane in a full arch custom tray. The models will be surveyed to produce CAD CAM crowns on RPD abutments which will incorporate design elements such as heights of contour and rest seats. Once cemented and following cast removable partial denture insertion, patients will be followed every year up for 3-5 years to assess outcomes.

Data Collection:

Independent Variables: Variables to be collected will include demographic data, age, sex and smoking status. Abutment tooth, reason for crown (including endodontic treatment, large restoration, replacement crown, change of axial morphology, tooth sensitivity), pulp vitality, history of previous endodontic treatment, presence of post core if any, type of core, status of opposing tooth whether present or absent or opposed by removable or fixed prosthesis, presence or absence of proximal contacts and type of cement used at insertion. Post insertion variables will include any and all follow up dates, and procedures performed at follow up.

Statistical Analysis: Descriptive statistics will be used to summarize patient characteristics and outcomes. For categorical variables, the investigators will report frequency and percentages. Numerical variables will be summarized using mean, standard deviation (or median/IQR for skewed distributions). For primary clinical outcomes, the investigators will also report 95% confidence intervals.

Sample size permitting, the investigators may also examine the association between baseline/demographic patient characteristics and outcomes using inferential analysis (chi-square tests, logistic/linear regression models). A level of significance 0.05 will be used for inferential analysis, with p-values < 0.05 reported as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: Patient recruitment will be from the adult patient population that presents to the undergraduate/graduate prosthodontic dental clinic requiring new tooth or tissue supported removable cast dental prostheses to replace missing teeth for the following situations:

  * In Kennedy Class 1 and 2 tisuue supported RPD's-Terminal abutments 3,4,5,6
  * In Kennedy Class 3 and 4 tooth supported RPD's- any abutment teeth selected will need to be documented if selected as abutments for a surveyed crown.
  * Selection of abutment teeth for zirconia surveyed crowns will be similar to that currently utilized when selecting cast RPD abutments to be restored with either porcelain fused to metal or full metal surveyed crowns for tissue and tooth supported cast RPD's. Identifiable data will include:
  * RPD abutment teeth which may benefit from full coverage due to large restorations.
  * Posterior endodontically treated teeth with inadequate marginal ridge support and
  * Abutment teeth which require axial modification for RPD retentive and or stability elements.
  * In situations where esthetic improvement is desirable
  * Reasons for selection wil be documented.

Exclusion Criteria:

* Crowns that need to be splinted; patients that decline a surveyed crown; patients under the age of 18 years; patients that decline to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2026-12-18 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | study follow up- every year for 3-5 years
  A. Survival will be recorded as the tooth with the crown still in function with or without 'clinical complications' during and up to the end of follow up. These will include but are not limited to
  * occlusal adjustments,
  * follow up sensitivity,
  * open margins,
  * recurrent decay,
  * infection,
  * endodontic treatment or retreatment,
  * chipping of ceramic,
  * recementation,
  * non healing endodontic lesion,
  * bone loss and associated periodontal problems.
Biological Complications | study follow up- every year for 3-5 years
  Biological failures will be recorded when the tooth is no longer present in the mouth either because of
  * tooth or core fracture rendering the tooth non restorable,
  * or the tooth extracted because of caries, infection or periodontal disease.
Technical Complications | study follow up- every year for 3-5 years
  Technical failures will be recorded when
  * the zirconia crown fractures or
  * needs to be replaced because of inadequate fit.
Success | study follow up- every year for 3-5 years
  Success will be recorded as all surviving crowns with no clinical complications.
Other complications | study follow up- every year for 3-5 years
  Not listed above

CONTACTS AND LOCATIONS:
Overall Officials: Eszter S Ganss, DDS, Study Chair — Faculty of Dentistry, University of Toronto

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be stored on secure university of Toronto servers and will be available only to researchers involved in the project

REFERENCES:
- [Background] Kois DE, Isvilanonda V, Chaiyabutr Y, Kois JC. Evaluation of fracture resistance and failure risks of posterior partial coverage restorations. J Esthet Restor Dent. 2013 Apr;25(2):110-22. doi: 10.1111/jerd.12018. Epub 2013 Mar 19. PMID 23617385
- [Background] Goto M, Oki K, Koyano K, Ayukawa Y. The 3-year cumulative survival rates of posterior monolithic zirconia crowns and their antagonist teeth, and their influencing factors. J Oral Sci. 2022 Oct 1;64(4):286-289. doi: 10.2334/josnusd.22-0221. Epub 2022 Sep 14. PMID 36104182
- [Background] Burns DR, Unger JW. The construction of crowns for removable partial denture abutment teeth. Quintessence Int. 1994 Jul;25(7):471-5. PMID 7991768
- [Background] Turner CH, Smith BJ. The use of crowns to modify abutment teeth of removable partial dentures. 2. Clinical and laboratory procedures. J Dent. 1979 Jun;7(2):98-104. doi: 10.1016/0300-5712(79)90002-2. No abstract available. PMID 379070
- [Background] Behr M, Kolbeck C, Lang R, Hahnel S, Dirschl L, Handel G. Clinical performance of cements as luting agents for telescopic double crown-retained removable partial and complete overdentures. Int J Prosthodont. 2009 Sep-Oct;22(5):479-87. PMID 20095198
- [Background] Kopzon V, Raedel M. Outcomes of abutment teeth with double crowns over an observation period of 27 years. J Prosthodont Res. 2023 Oct 13;67(4):518-523. doi: 10.2186/jpr.JPR_D_22_00165. Epub 2022 Dec 17. PMID 36529501
- [Background] Igarashi Y, Goto T. Ten-year follow-up study of conical crown-retained dentures. Int J Prosthodont. 1997 Mar-Apr;10(2):149-55. PMID 9206455
- [Background] Sorensen JA, Martinoff JT. Endodontically treated teeth as abutments. J Prosthet Dent. 1985 May;53(5):631-6. doi: 10.1016/0022-3913(85)90008-3. No abstract available. PMID 3889302
- [Background] D'Souza NL, Jutlah EM, Deshpande RA, Somogyi-Ganss E. Comparison of clinical outcomes between single metal-ceramic and zirconia crowns. J Prosthet Dent. 2025 Feb;133(2):464-471. doi: 10.1016/j.prosdent.2024.02.028. Epub 2024 Apr 4. PMID 38580582